CLINICAL TRIAL: NCT04852575
Title: ReVital Chemotherapy Online Resiliency Evaluation (ReVital-CORE) Program Pilot Feasibility Study
Brief Title: ReVital-CORE Program
Acronym: ReVital-CORE
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Collaborators: Select Medical (Unknown)
Responsible Party: Principal Investigator, Mackenzi Pergolotti, Senior Director, Research and Clinical Development, Kessler Foundation
Other Study IDs: E-1132-20
Record Dates: First submitted 2021-03-01; First posted 2021-04-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Frailty; Cancer; Chemotherapy-Induced Change
Keywords: Frailty; Cancer; Chemotherapy; Care coordination; Online; Prospective surveillance
MeSH Terms: conditions — Frailty; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pilot feasibility study of the ReVital Chemotherapy Online Resiliency Evaluation (CORE) program. As part of standard of care, patients starting a new chemotherapy regimen are referred to complete a pre-chemotherapy cancer rehabilitation evaluation (i.e., prehab) and invited to enroll in the ReVital-CORE program study.

Once enrolled in ReVital-CORE, participants will complete a monthly online evaluation for 1 year. If frailty (or pre-frailty) is detected on any survey, physical or occupational therapy will be initiated for standard of care rehabilitation evaluation and treatment.

DETAILED DESCRIPTION:
All patients starting a new chemotherapy regimen will be referred to completed a prehab evaluation with a specialized physical or occupational therapist be and invited to enroll in the ReVital-CORE program for the pilot, feasibility study.

Participants in the ReVital-CORE program study will be emailed an online evaluation each month via for one year. Once completed, the evaluation is automatically scored into: frail, pre-frail or robust categories using a validated frailty index. Any patient categorized as frail or pre-frail will be re-referred to rehabilitation by their cancer care team. For frail and pre-frail individuals, standard of care rehabilitation therapy will include either/and occupational and physical therapy evaluation and treatment and will be billed via their insurance.

The purpose of this pilot study is to evaluate feasibility of the of the ReVital-CORE Program for individuals starting a new chemotherapy regimen. Secondary aims are to evaluate the prevalence, trajectory and predictors of frailty during the first year of chemotherapy treatment; and evaluate the impacts of prehab/rehabilitation for participants identified as frail and pre-frail.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* English speaking
* Starting new chemotherapy treatment with oncology partner
* Provide informed consent

Exclusion Criteria:

* Eligible for hospice care

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with cancer who are starting a new chemotherapy regimen (note: can be any line of chemotherapy)
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Accrual to the ReVital-CORE program. | 02/2022
  Proportion of patients who consent to enroll, out of the total number invited.

SECONDARY OUTCOMES:
Prevalence of frailty at major time points. | 02/2023
  Proportion of participants at all major timepoints (pre-chemo, and monthly following start of chemo for 12 months) who are identified as frail or pre-frail by a patient-reported frailty index.
Impact of therapy on global quality of life. | 02/2023
  Change from baseline to discharge in quality of life as measured by the Patient Reported Outcomes Measuring System (PROMIS)-global 10-item questionnaire.
Impact of therapy on frailty. | 02/2023
  Change from baseline to discharge in frailty as measured by a patient-reported frailty index.

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzi Pergolotti, PhD, Principal Investigator — Select Medical
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.